CLINICAL TRIAL: NCT05618314
Title: A Phase 1, Open-Label, Parallel-Group, Single-Dose Adaptive Study to Evaluate the Safety and Pharmacokinetics of AT-527 in Adult Subjects With Normal and Impaired Renal Function Sub-Study: Effects of Probenecid on the Pharmacokinetics of AT-527 in Healthy Adult Subjects
Brief Title: Study of AT-527 in Subjects With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-011
Record Dates: First submitted 2022-10-26; First posted 2022-11-16 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteer; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — AT-511; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group A-Mild Renal Impairment (Experimental): single dose AT-527
  Interventions: Drug: AT-527
- Group B-Moderate Renal Impairment (Experimental): single dose AT-527
  Interventions: Drug: AT-527
- Group C-Severe Renal Impairment (optional) (Experimental): single dose AT-527
  Interventions: Drug: AT-527
- Group D-End-Stage Renal Disease (optional) (Experimental): single dose of AT-527 pre- and post-dialysis
  Interventions: Drug: AT-527
- Group E-Matched Healthy Subjects (Experimental): Single dose of AT-527 on Days 1 and 15. Probenecid administered twice daily (BID) Days 14-19
  Interventions: Drug: AT-527 and Probenecid

INTERVENTIONS:
Drug: AT-527 — single dose AT-527
  Other Names: Bemnifosbuvir
  Arms: Group A-Mild Renal Impairment; Group B-Moderate Renal Impairment; Group C-Severe Renal Impairment (optional)
Drug: AT-527 — Single dose of AT-527 pre- and post-dialysis
  Other Names: Bemnifosbuvir
  Arms: Group D-End-Stage Renal Disease (optional)
Drug: AT-527 and Probenecid — Single dose of AT-527 on Days 1 and 15. Probenecid administered twice daily (BID) Days 14-19
  Other Names: Bemnifosbuvir
  Arms: Group E-Matched Healthy Subjects

SUMMARY:
Study of AT-527 in Subjects with Normal and Impaired Renal Function

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* BMI of 18.5 to 42.0 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Subjects with Normal Renal Function (Group E):

* Medically healthy, in the opinion of an Investigator
* Normal renal function with eGFR ≥ 90 mL/min/1.73m2 at Screening

Renal Impaired Subjects (Groups A, B, and C):

* Considered stable in the judgement of an Investigator
* Presence of severe renal impairment (eGFR ≥ 15 and < 30 mL/min/1.73m2), moderate renal impairment (eGFR ≥ 30 and < 60 mL/min/1.73m2) or mild renal impairment (eGFR ≥ 60 and < 90 mL/min/1.73m2) at Screening: renal impairment should have been stable for at least 1 month prior to Screening.

Subjects with End-Stage Renal Disease -ESRD (Group D)

* Considered clinically stable in the opinion of the Investigator
* Presence of ESRD (eGFR <15 mL/min/1.73m2 and being on intermittent hemodialysis) at Screening and have been stable for at least 1 month prior to Screening

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with HIV or COVID-19
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Subjects with Normal Renal Function (Group E):

• Any clinically significant illness in the opinion of the investigator

Subjects with Impaired Renal Function (Group A, B, C and D):

* History of renal transplant
* Presence of poorly controlled Type 1 or Type 2 diabetes as defined by Hemoglobin A1c (HbA1c) > 10%
* Subjects requiring treatment for renal impairment or other chronic disease must be on a stable treatment plan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of AT-527 Maximum plasma concentration (Cmax) | Day 1
Pharmacokinetics (PK) of AT-527 Area under the plasma concentration-time curve (AUC) | Day 1
Pharmacokinetics (PK) of AT-527 AUC | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Québec, Canada

IPD SHARING:
Plan to Share IPD: No